CLINICAL TRIAL: NCT00418561
Title: A Single Center, Open-label, Non-randomized, Uncontrolled, Multiple-dose, Dose Escalation Study of the Safety, Pharmacokinetics and Efficacy of Metazym for the Treatment of Patients With Late Infantile Metachromatic Leukodystrophy (MLD)
Brief Title: Metazym for the Treatment of Patients With Late Infantile Metachromatic Leukodystrophy (MLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: rhASA-01; 2006-005341-11 (EudraCT Number)
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Metachromatic Leukodystrophy (MLD)
Keywords: rhASA; MLD; Metazym
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Metazym (Recombinant human arylsulfatase A (rhASA)): 25 U/kg as a single dose - hereafter 50 U/kg
  Interventions: Biological: rhASA - Dose Level 1
- Cohort 2 (Experimental): 100 U/kg Metazym (Recombinant human arylsulfatase A (rhASA))
  Interventions: Biological: rhASA - Dose Level 2
- Cohort 3 (Experimental): 200 U/kg Metazym (Recombinant human arylsulfatase A (rhASA))
  Interventions: Biological: rhASA - Dose Level 3

INTERVENTIONS:
Biological: rhASA - Dose Level 1 — Intravenous infusion 25 U/kg as a single dose - hereafter 50 U/kg every other week for 26 weeks
  Other Names: HGT-1111; metazym
  Arms: Cohort 1
Biological: rhASA - Dose Level 2 — Intravenous infusion 100 U/kg every other week for 26 weeks
  Other Names: HGT-1111; metazym
  Arms: Cohort 2
Biological: rhASA - Dose Level 3 — Intravenous infusion 200 U/kg every other week for 26 weeks
  Other Names: HGT-1111; metazym
  Arms: Cohort 3

SUMMARY:
Objectives: The overall objective is to evaluate the safety, efficacy and pharmacokinetics (PK) of rhASA treatment in patients with late infantile MLD.

Methodology: This is a single center, open-label study of patients with late infantile MLD. Twelve patients will be enrolled in this study receiving a total of thirteen intravenous infusions of Metazym. One infusion will be given every other week for a period of half a year. After the half year the subjects will continue treatment every other week until safety data is available. Safety (AE/SAE) will be monitored at every visit during this period.

DETAILED DESCRIPTION:
Test product, dose, mode of administration, batch No.: The lowest dose level will be evaluated as a single dose of 25 U/kg. The three upper dose levels will be evaluated as repeated doses. Patients in each cohort will receive one dose of enzyme every other week for a period of eight weeks, a total of five doses. Dosing will be performed as follows: Cohort 1: 25 U/kg as a single dose - hereafter 50 U/kg; Cohort 2: 100 U/kg; Cohort 3: 200 U/kg. Patients receiving the lowest dose as a single dose will receive the next dose level as a repeated dose. After twenty six weeks the subjects will continue treatment every other week until safety data is available. Safety (AE/SAE) will be monitored at every visit during this period. The dose will be adjusted monthly to account for changes in body weight. The infusion length will be dependent on the dose. Doses of 25 U/kg, 50 U/kg and 100 U/kg will be diluted in 50 ml isotonic sodium chloride and infused over 30 minutes. Infusion of 200 U/kg will be administered in the same manner except for an infusion time of 60 minutes.

Duration of treatment: Half a year (26 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. Subject's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities (Trial-related activities are any procedures that would not have been performed during normal management of the subject).
2. The patient must have a confirmed diagnosis of MLD as defined by:

   ASA activity < 10 nmol/h/mg in leukocytes Presence of elevated sulfatide in urine
3. The patient must have a confirmed nerve conduction velocity < 2 standard deviations (from the appropriate age level)
4. The patient must have a residual level of voluntary function (as judged by the investigator), including presence of residual cognitive function (attention, executive and visual functions) as well as the presence of residual voluntary motor function in one upper or lower limb as a minimum.
5. The patient must have an age at the time of screening ≥ 1 year and < 6 years
6. The patient must have had onset of symptoms before the age of 4 years
7. The subject and his/her guardian(s) must have the ability to comply with the clinical protocol
8. The patients' medical record must document that the legal guardian(s) has had independent counselling or a consultation regarding stem cell transplantation in order to assure that the guardian(s) is fully informed regarding the risks and benefits of this alternative

Exclusion Criteria:

Patients will be excluded from this study if they do not meet the specific inclusion criteria, or if any of the following criteria apply:

1. Lack of voluntary function
2. Presence of severe pseudo-bulbar signs (weakness and disco-ordination of tongue and swallowing muscles leading to severe difficulty with swallowing)
3. Spasticity so severe to inhibit transportation
4. Known multiple sulfatase deficiency
5. Presence of major congenital abnormality
6. Presence of known chromosomal abnormality and syndromes affecting psychomotor development
7. History of stem cell transplantation
8. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition
9. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial
10. Use of any investigational product within 30 days prior to study enrolment or currently enrolled in another study which involves clinical investigations
11. Received ERT with rhASA from any source
12. Planned or anticipated initiation of antispastic treatment after trial initiation

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2008-03-27 (Actual); Study Completion 2008-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Rigshospitalet, Hvidovre, Denmark

REFERENCES:
- [Result] Dali CI, Barton NW, Farah MH, Moldovan M, Mansson JE, Nair N, Duno M, Risom L, Cao H, Pan L, Sellos-Moura M, Corse AM, Krarup C. Sulfatide levels correlate with severity of neuropathy in metachromatic leukodystrophy. Ann Clin Transl Neurol. 2015 May;2(5):518-33. doi: 10.1002/acn3.193. Epub 2015 Mar 27. PMID 26000324
- [Derived] I Dali C, Groeschel S, Moldovan M, Farah MH, Krageloh-Mann I, Wasilewski M, Li J, Barton N, Krarup C. Intravenous arylsulfatase A in metachromatic leukodystrophy: a phase 1/2 study. Ann Clin Transl Neurol. 2021 Jan;8(1):66-80. doi: 10.1002/acn3.51254. Epub 2020 Dec 17. PMID 33332761

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Single dose of 25 U/kg recombinant human Arylsulphatase A (Metazym, rhASA), thereafter, received repeated doses of 50 U/kg recombinant human Arylsulphatase A, once in every 2 weeks for a period of 26 weeks, as an intravenous (IV) infusion over 30 minutes. Dosage adjustment was done monthly to account for changes in body weight.
- Cohort 2: Repeated doses of 100 U/kg recombinant human Arylsulphatase A (Metazym, rhASA), once in every 2 weeks for a period of 26 weeks, as an IV infusion over 30 minutes. Dosage adjustment was done monthly to account for changes in body weight.
- Cohort 3: Repeated doses of 200 U/kg recombinant human Arylsulphatase A (Metazym, rhASA), once in every 2 weeks for a period of 26 weeks, as an IV infusion over 60 minutes. Dosage adjustment was done monthly to account for changes in body weight.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 4 | 5 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 1 | 0
Not completed — Participant's (guardian's) decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: Single dose of 25 U/kg recombinant human Arylsulphatase A (Metazym, rhASA), thereafter, received repeated doses of 50 U/kg recombinant human Arylsulphatase A, once in every 2 weeks for a period of 26 weeks, as an IV infusion over 30 minutes. Dosage adjustment was done monthly to account for changes in body weight.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: months] | 36.25 (9.32) | 41.80 (10.13) | 30.75 (7.27) | 36.69 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurring in a participant, participating in a clinical study with study drug, regardless of causal relationship. TEAEs were AEs occurred after study drug administration that were absent before treatment or that worsened relative to pre-treatment state, up to Week 28 until evaluation (when last cohort had 26-week evaluation and data management performed within 4 weeks) completed.
Time Frame: From study drug administration up to Week 28
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
participants | 4 | 5 | 4

2. Primary Outcome: Change From Baseline in Gross Motor Function Measure (GMFM) at Week 26
Description: GMFM was measured using GMFM-88 item scores and summed to calculate a total GMFM-88 score. For each GMFM-88 item, the score was between 0 (minimal) to 3 (maximum). The total GMFM-88 score was between 0 (minimal) and 264 (maximum). The decrease in GMFM score over time indicates worsening of disease over time. Relative change from baseline at Week 26 was calculated as percentage change from baseline divided by the age-difference in months between first and last visit. Adjusted mean and 95 percent (%) confidence intervals were reported.
Time Frame: Baseline, Week 26
Population: ITT
Measure: Mean (95% Confidence Interval); unit: percent (%) change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
percent (%) change | -2.36 [-7.62 to 2.91] | -8.29 [-13.55 to -3.02] | -10.90 [-16.17 to -5.64]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; The comparisons of the three doses were done using analysis of variance (ANOVA) model including the baseline measurement as a covariate; Test type: Superiority or Other; p = 0.0737, ANOVA — Test for no difference between cohorts

3. Primary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Sulfatide at Week 26
Description: Relative change from baseline at Week 26 was calculated as percentage change from baseline divided by the age-difference in months between first and last visit. Adjusted mean and 95 percent (%) confidence intervals were reported.
Time Frame: Baseline, Week 26
Population: ITT
Measure: Mean (95% Confidence Interval); unit: percent (%) change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
percent (%) change | 24.55 [0.44 to 48.66] | -3.77 [-22.33 to 14.80] | -4.32 [-28.17 to 19.53]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; The comparisons of the three doses were done using ANOVA model including the baseline measurement as a covariate; Test type: Superiority or Other; p = 0.1115, ANOVA — Test for no difference between cohorts

4. Primary Outcome: Number of Participants With Shift From Baseline to Week 26 in Sulfatide Levels in Urine
Description: Number of participants with shifts between negative (value=0) and positive (value=1) values in urine sulfatide levels from baseline at Week 26 is reported.
Time Frame: Baseline up to Week 26
Population: ITT. Here, the number of participants analyzed are the participants evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 2 | 2
participants
  Negative(0) to negative(0) | 0 | 0 | 0
  Negative(0) to positive(1) | 0 | 0 | 0
  Positive(1) to negative(0) | 0 | 0 | 0
  Positive(1) to positive(1) | 3 | 2 | 2

5. Primary Outcome: Change From Baseline in Mullen's Scales of Early Learning at Week 26
Description: Mullen's Scales of Early Learning is used to assess performance and learning ability in young children. The scale consisted of 144 items that had specific scoring criteria for each item. The scores were converted to T-scores with a decrease in score indicating worsening of disease. Relative change from baseline at Week 26 was calculated as percentage change from baseline divided by the age-difference in months between first and last visit. Adjusted mean and 95 percent (%) confidence intervals were reported.
Time Frame: Baseline, Week 26
Population: ITT
Measure: Mean (95% Confidence Interval); unit: percent (%) change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
percent (%) change | 16.28 [0.72 to 31.84] | 0.26 [-15.49 to 16.02] | -4.92 [-20.26 to 10.41]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; The comparisons of the three doses were done using ANOVA model including the baseline measurement as a covariate; Test type: Superiority or Other; p = 0.1268, ANOVA — Test for no difference between cohorts

6. Secondary Outcome: Change From Baseline in Nerve Conduction Velocity at Week 26
Description: An electrophysiological evaluation using standard electrophysiological and electromyography to measure the speed and extent of nerve conduction and units are expressed in meters per second. Abbreviations: MN=Median Nerve; PN=Peroneal Nerve; SN=Sural Nerve; Dig.=Digit; FH=fibular hemimelia; L LM=left lateral medial; R LM=right lateral medial; MC=medial collateral.
Time Frame: Baseline, Week 26
Population: ITT. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
meters per second
  MN, Elbow Wrist: Baseline (N=4,5,4) | 20.38 (6.99) | 25.78 (17.72) | 15.95 (5.68)
  MN, Elbow Wrist: Change at Week 26 (N=4,4,4) | -4.00 (1.10) | 2.62 (4.42) | -3.65 (3.33)
  MN, Dig. II Wrist: Baseline (N=3,5,4) | 39.83 (7.22) | 36.82 (16.64) | 23.30 (11.99)
  MN, Dig. II Wrist: Change at Week 26 (N=3,4,4) | -11.7 (5.78) | -0.25 (4.39) | -1.33 (4.72)
  PN, Dig. Ankle FH: Baseline (N=4,4,4) | 20.70 (9.08) | 32.23 (21.41) | 14.13 (5.92)
  PN, Dig. Ankle FH: Change at Week 26 (N=4,3,4) | -7.85 (3.92) | -2.43 (1.59) | -2.65 (3.61)
  SN, Sensory L LM - MC: Baseline (N=4,4,4) | 26.88 (9.29) | 36.13 (20.61) | 29.18 (15.93)
  SN, Sensory L LM - MC: Change at Week 26 (N=3,3,4) | -5.57 (4.18) | 3.70 (9.79) | -9.33 (10.64)
  SN, Sensory R LM - MC: Baseline (N=4,4,4) | 31.35 (6.46) | 34.58 (17.74) | 27.48 (13.91)
  SN, Sensory R LM - MC: Change at Week 26 (N=0,0,0) | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported. | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported. | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported.

7. Secondary Outcome: Number of Participants Who Had Undergone Nerve Biopsy and Had a Normal Nerve at Both Baseline and Week 26
Time Frame: Baseline, Week 26
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
participants
  Baseline | 0 | 2 | 0
  Week 26 | 0 | 2 | 0

8. Secondary Outcome: Number of Participants With Shift From Baseline to Week 26 in Magnetic Resonance Imaging (MRI)-Loes Scores
Description: Loes scoring system is used to grade the demyelinating abnormalities on brain MRI. A total of 17 locations of the brain were scored from 0 (normal appearance) to 2 (dense appearance). The total score ranged from 0 to 34 with a score of 14 or greater being considered severe. Number of participants with any shift of score between 0 to 2 for each of the 17 locations (Parieto Occipital [PO]-Periventricular [P], Central [C], Subcortical [Sc]; Anterior Temporal [AT]-P, C, Sc; Frontal [F]-P, C, Sc; Corpus Callosum [CC]-Splenium [S], Genus [G]; Projection Fibers [PF]-Capsular interna [CI] ant, CI post, Brainstem [B]; Cerebellum [Cb]-Cortex, Atrophy; Basal Ganglia [BG]-BG, Thalamus [T]; Cerebral Atrophy [CA]-CA), are only reported.
Time Frame: Baseline up to Week 26
Population: ITT. Here, number of participants analyzed in the Cohort 2 are the participants evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
participants
  PO, P: 1 to 2 | 1 | 0 | 1
  PO, P: 2 to 2 | 3 | 4 | 3
  PO, C: 2 to 2 | 4 | 4 | 4
  PO, Sc: 0 to 0 | 1 | 0 | 1
  PO, Sc: 0 to 1 | 0 | 1 | 0
  PO, Sc: 0 to 2 | 0 | 0 | 1
  PO, Sc: 1 to 1 | 0 | 1 | 0
  PO, Sc: 1 to 2 | 0 | 0 | 1
  PO, Sc: 2 to 2 | 3 | 2 | 1
  AT, P: 0 to 2 | 1 | 0 | 0
  AT, P: 1 to 2 | 0 | 1 | 2
  AT, P: 2 to 2 | 3 | 3 | 2
  AT, C: 0 to 2 | 1 | 0 | 0
  AT, C: 1 to 2 | 0 | 0 | 1
  AT, C: 2 to 2 | 3 | 4 | 3
  AT, Sc: 0 to 0 | 1 | 0 | 1
  AT, Sc: 0 to 1 | 0 | 1 | 0
  AT, Sc: 0 to 2 | 0 | 2 | 2
  AT, Sc: 1 to 1 | 0 | 1 | 0
  AT, Sc: 1 to 2 | 1 | 0 | 0
  AT, Sc: 2 to 2 | 2 | 0 | 1
  F, P: 0 to 2 | 1 | 0 | 1
  F, P: 1 to 2 | 0 | 1 | 1
  F, P: 2 to 2 | 3 | 3 | 2
  F, C: 1 to 2 | 1 | 0 | 2
  F, C: 2 to 2 | 3 | 4 | 2
  F, Sc: 0 to 0 | 1 | 0 | 1
  F, Sc: 0 to 2 | 0 | 2 | 2
  F, Sc: 1 to 2 | 1 | 1 | 0
  F, Sc: 2 to 2 | 2 | 1 | 1
  CC, S: 1 to 0 | 0 | 1 | 1
  CC, S: 1 to 2 | 1 | 0 | 0
  CC, S: 2 to 0 | 1 | 1 | 1
  CC, S: 2 to 1 | 2 | 1 | 0
  CC, S: 2 to 2 | 0 | 1 | 2
  CC, G: 0 to 2 | 1 | 1 | 0
  CC, G: 1 to 1 | 0 | 1 | 0
  CC, G: 1 to 2 | 0 | 0 | 2
  CC, G: 2 to 1 | 1 | 0 | 1
  CC, G: 2 to 2 | 2 | 2 | 1
  PF, CI ant: 0 to 0 | 2 | 3 | 4
  PF, CI ant: 0 to 1 | 1 | 1 | 0
  PF, CI ant: 1 to 1 | 1 | 0 | 0
  PF, CI post: 0 to 0 | 0 | 1 | 0
  PF, CI post: 0 to 1 | 1 | 0 | 2
  PF, CI post: 1 to 1 | 0 | 2 | 0
  PF, CI post: 1 to 2 | 1 | 0 | 1
  PF, CI post: 2 to 1 | 0 | 1 | 0
  PF, CI post: 2 to 2 | 2 | 0 | 1
  PF, B: 0 to 0 | 1 | 0 | 1
  PF, B: 0 to 1 | 0 | 1 | 1
  PF, B: 0 to 2 | 0 | 0 | 1
  PF, B: 1 to 0 | 0 | 1 | 0
  PF, B: 1 to 1 | 1 | 0 | 0
  PF, B: 1 to 2 | 1 | 1 | 1
  PF, B: 2 to 2 | 1 | 1 | 0
  Cb, Cortex: 0 to 0 | 2 | 1 | 1
  Cb, Cortex: 0 to 1 | 0 | 2 | 2
  Cb, Cortex: 1 to 1 | 2 | 1 | 1
  Cb, Atrophy: 0 to 0 | 1 | 1 | 3
  Cb, Atrophy: 0 to 1 | 1 | 1 | 0
  Cb, Atrophy: 1 to 1 | 2 | 2 | 1
  Bg, Bg: 0 to 0 | 2 | 3 | 2
  Bg, Bg: 0 to 1 | 0 | 0 | 2
  Bg, Bg: 1 to 0 | 0 | 1 | 0
  Bg, Bg: 1 to 1 | 2 | 0 | 0
  Bg, T: 0 to 0 | 2 | 3 | 3
  Bg, T: 1 to 0 | 0 | 1 | 1
  Bg, T: 1 to 1 | 2 | 0 | 0
  CA, CA: 0 to 0 | 1 | 0 | 2
  CA, CA: 0 to 1 | 0 | 2 | 1
  CA, CA: 1 to 1 | 1 | 1 | 1
  CA, CA: 1 to 2 | 2 | 1 | 0

9. Secondary Outcome: Change From Baseline in Paediatric Evaluation of Disability Inventory (PEDI) Scores at Week 26
Description: PEDI is used for the clinical evaluation of functional capabilities, performance and changes in functional skills in children with disabilities. It consisted of 20 items scored on a scale from 0 (total assistance) to 5 (independent). Total score ranged from 0-100 with higher scores indicating better functioning. None, child, rehab, extensive are items in 3 domains (self-care, mobility and social functioning).
Time Frame: Baseline, Week 26
Population: ITT. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
units on a scale
  Self-care, None: Baseline (N=4,5,4) | 6.25 (0.96) | 6.00 (1.41) | 4.75 (2.06)
  Self-care, None: Change at Week 26 (N=4,4,4) | -0.75 (1.50) | -1.50 (1.73) | -1.50 (1.91)
  Self-care, Child: Baseline (N=4,5,4) | 1.75 (0.96) | 2.00 (1.41) | 3.25 (2.06)
  Self-care, Child: Change at Week 26 (N=4,4,4) | 0.75 (1.50) | 1.25 (1.50) | 0.75 (2.22)
  Self-care, Rehab: Baseline (N=4,5,4) | 0 (0) | 0 (0) | 0 (0)
  Self-care, Rehab: Change at Week 26 (N=4,4,4) | 0 (0) | 0 (0) | 0 (0)
  Self-care, Extensive: Baseline (N=4,5,4) | 0 (0) | 0.20 (0.45) | 0 (0)
  Self-care, Extensive: Change at Week 26 (N=4,4,4) | 0 (0) | 0.25 (0.50) | 0.50 (0.58)
  Mobility, None: Baseline (N=4,5,4) | 4.25 (1.89) | 3.60 (1.14) | 5.00 (0.82)
  Mobility, None: Change at Week 26 (N=4,4,4) | -0.75 (1.71) | -0.50 (1.29) | -1.25 (1.71)
  Mobility, Child: Baseline (N=4,5,4) | 2.50 (1.91) | 2.40 (1.67) | 1.25 (1.26)
  Mobility, Child: Change at Week 26 (N=4,4,4) | 0.00 (1.41) | 0.25 (1.26) | -0.50 (0.58)
  Mobility, Rehab: Baseline (N=4,5,4) | 0.00 (0.00) | 1.00 (1.41) | 0.75 (0.96)
  Mobility, Rehab: Change at Week 26 (N=4,4,4) | 1.00 (0.82) | 0.25 (0.50) | 0.50 (1.73)
  Mobility, Extensive: Baseline (N=4,5,4) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Mobility, Extensive: Change at Week 26 (N=4,4,4) | 0.00 (0.00) | 0.00 (0.00) | 1.25 (1.50)
  Social, None: Baseline (N=4,5,4) | 4.25 (0.96) | 4.60 (0.55) | 4.75 (0.50)
  Social, None: Change at Week 26 (N=4,4,4) | 0.75 (0.96) | -0.25 (0.50) | 0.25 (0.50)
  Social, Child: Baseline (N=4,5,4) | 1.50 (2.38) | 0.00 (0.00) | 0.25 (0.50)
  Social, Child: Change at Week 26 (N=4,4,4) | -1.50 (2.38) | 0.00 (0.00) | -0.25 (0.50)
  Social, Rehab: Baseline (N=4,5,4) | 0.00 (0.00) | 0.40 (0.55) | 0.00 (0.00)
  Social, Rehab: Change at Week 26 (N=4,4,4) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Social, Extensive: Baseline (N=4,5,4) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Social, Extensive: Change at Week 26 (N=4,4,4) | 0.00 (0.00) | 0.25 (0.50) | 0.00 (0.00)

10. Other Pre Specified Outcome: Number of Participants With Shift From Baseline to Week 26 in Clinical Laboratory Evaluations: Biochemistry
Description: Number of participants with at least 1 shift from baseline to Week 26, are reported. Abbreviations: ALT=Alanine transaminase; CK=Creatine kinase; AP=Amyloid P component; LDH=Lactate dehydrogenase.
Time Frame: Baseline up to Week 26
Population: ITT. Here, number of participants analyzed in the Cohort 2 are the participants evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
participants
  ALT-Serum: Low to low | 2 | 0 | 1
  ALT-Serum: Low to normal | 1 | 1 | 0
  ALT-Serum: Normal to low | 0 | 1 | 2
  ALT-Serum: Normal to normal | 0 | 1 | 1
  ALT-Serum: High to low | 1 | 0 | 0
  ALT-Serum: High to normal | 0 | 1 | 0
  Amylase-Serum: Normal to normal | 4 | 4 | 4
  AP-Serum: Normal to normal | 4 | 4 | 4
  Calcium-Serum: Normal to normal | 4 | 3 | 4
  CK-Serum: Normal to normal | 4 | 3 | 2
  CK-Serum: Normal to high | 0 | 1 | 0
  CK-Serum: High to normal | 0 | 0 | 1
  CK-Serum: High to high | 0 | 0 | 1
  Creatinine-Serum: Normal to normal | 4 | 4 | 4
  Iron-Serum: Low to normal | 0 | 1 | 0
  Iron-Serum: Normal to low | 0 | 0 | 1
  Iron-Serum: Normal to normal | 3 | 3 | 3
  Iron-Serum: Normal to high | 1 | 0 | 0
  LDH-Serum: Normal to normal | 3 | 4 | 4
  LDH-Serum: High to normal | 1 | 0 | 0
  Magnesium-Serum: Normal to normal | 4 | 4 | 4
  Phosphate-Serum: Normal to normal | 2 | 3 | 3
  Phosphate-Serum: Normal to high | 1 | 0 | 0
  Phosphate-Serum: High to normal | 1 | 1 | 1
  Potassium-Serum: Normal to normal | 4 | 4 | 4
  Sodium-Serum: Normal to normal | 4 | 3 | 4
  Sodium-Serum: High to normal | 0 | 1 | 0
  T Bilirubin-Serum: Normal to normal | 4 | 3 | 4
  T Bilirubin-Serum: High to normal | 0 | 1 | 0

11. Other Pre Specified Outcome: Number of Participants With Shift From Baseline to Week 26 in Clinical Laboratory Evaluations: Coagulation
Description: Number of participants with at least 1 shift from baseline to Week 26 are reported. The shift reported below for Cohort 1 was from low level at baseline to low level at Week 26.
Time Frame: Baseline up to Week 26
Population: ITT. Data for Cohorts 2 and 3 were not reported since there were no participants with shift from baseline to Week 26 in coagulation evaluations.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 0 | 0
participants | 4 |  |

12. Other Pre Specified Outcome: Number of Participants With Shift From Baseline to Week 26 in Clinical Laboratory Evaluations: Genotyping
Description: Number of participants with at least 1 shift from baseline to Week 26 are reported. Abbreviations: CSF=Cerebrospinal fluid; NFP=Neurofilament proteins.
Time Frame: Baseline up to Week 26
Population: ITT. The number of participants analyzed in the Cohort 2 are the participants evaluable for this outcome. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
participants
  Albumin CSF: Normal to normal (N=3,4,4) | 0 | 2 | 0
  Albumin CSF: Normal to high (N=3,4,4) | 1 | 0 | 0
  Albumin CSF: High to high (N=3,4,4) | 2 | 2 | 4
  Albumin index: Normal to normal (N=3,4,4) | 0 | 1 | 0
  Albumin index: High to high (N=3,4,4) | 3 | 3 | 4
  Albumin Serum: Low to low (N=3,4,4) | 2 | 2 | 2
  Albumin Serum: Low to normal (N=3,4,4) | 0 | 1 | 0
  Albumin Serum: Normal to low (N=3,4,4) | 0 | 0 | 1
  Albumin Serum: Normal to normal (N=3,4,4) | 1 | 1 | 1
  Chitotriosidase CSF: Low to low (N=4,4,4) | 1 | 0 | 0
  Chitotriosidase CSF: High to high (N=4,4,4) | 3 | 4 | 4
  NFP CSF: Normal to high (N=4,4,4) | 1 | 0 | 0
  NFP CSF: High to high (N=4,4,4) | 3 | 4 | 4
  Sulfatide CSF: High to high (N=3,4,4) | 3 | 4 | 4
  Tauprotein CSF: High to low (N=4,4,4) | 0 | 1 | 0
  Tauprotein CSF: High to high (N=4,4,4) | 4 | 3 | 4

13. Other Pre Specified Outcome: Number of Participants With Shift From Baseline to Week 26 in Clinical Laboratory Evaluations: Hematology
Description: Number of participants with at least 1 shift from baseline to Week 26 are reported. Abbreviations: Abs=Absolute count; ERCS=Erythrocytes; MCHC=Mean corpuscular hemoglobin concentration; MCH=Mean cell hemoglobin.
Time Frame: Baseline up to Week 26
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 4 | 4
participants
  Basophils Abs - Blood: Normal to normal (N=4,4,4) | 4 | 4 | 4
  Eosinophil Abs - Blood: Normal to normal (N=4,4,4) | 4 | 4 | 4
  ERCS - Blood: Low to low (N=4,4,4) | 1 | 0 | 0
  ERCS - Blood: Normal to normal (N=4,4,4) | 3 | 4 | 4
  Haemoglobin - Blood: Low to low (N=4,4,4) | 1 | 1 | 1
  Haemoglobin - Blood: Low to normal (N=4,4,4) | 1 | 0 | 1
  Haemoglobin - Blood: Normal to low (N=4,4,4) | 1 | 0 | 1
  Haemoglobin - Blood: Normal to normal (N=4,4,4) | 1 | 3 | 1
  Lymphocyte Abs - Blood: Low to low (N=4,4,4) | 0 | 1 | 0
  Lymphocyte Abs - Blood: Normal to low (N=4,4,4) | 2 | 2 | 2
  Lymphocyte Abs - Blood: Normal to normal (N=4,4,4) | 2 | 1 | 2
  MCHC - Blood: Normal to normal (N=4,4,4) | 3 | 3 | 4
  MCHC - Blood: High to normal (N=4,4,4) | 1 | 1 | 0
  MCH - Blood: Low to low (N=4,4,4) | 0 | 0 | 1
  MCH - Blood: Normal to normal (N=4,4,4) | 4 | 4 | 3
  Monocytes Abs - Blood: Normal to normal (N=4,4,4) | 4 | 4 | 3
  Monocytes Abs - Blood: High to normal (N=4,4,4) | 0 | 0 | 1
  Neutropil Abs - Blood: Normal to normal (N=4,4,4) | 4 | 4 | 3
  Neutropil Abs - Blood: Normal to high (N=4,4,4) | 0 | 0 | 1
  Thrombocytes - Blood: Normal to low (N=4,3,4) | 1 | 0 | 1
  Thrombocytes - Blood: Normal to normal (N=4,3,4) | 2 | 0 | 2
  Thrombocytes - Blood: High to normal (N=4,3,4) | 1 | 3 | 1
  T Leucocytes - Blood: Low to normal (N=4,4,4) | 0 | 0 | 1
  T Leucocytes - Blood: Normal to low (N=4,4,4) | 2 | 2 | 0
  T Leucocytes - Blood: Normal to normal (N=4,4,4) | 2 | 2 | 3

14. Other Pre Specified Outcome: Number of Participants With Abnormal Findings in Urine Analysis
Description: The parameters analyzed in urine were albumin/protein, glucose, leucocytes, acetoacetate/ketones, nitrite and pH. Urine analysis findings were considered abnormal as judged by the investigator.
Time Frame: Baseline up to Week 26
Population: ITT
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
participants | 0 | 0 | 0

15. Other Pre Specified Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: Abnormal ECG findings were considered as clinically significant at the discretion of investigator.
Time Frame: Baseline up to Week 26
Population: ITT
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
participants | 0 | 0 | 0

16. Other Pre Specified Outcome: Change From Baseline in Chitotriosidase at Week 26
Time Frame: Baseline, Week 26
Population: ITT. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Mean (Standard Deviation); unit: nanomole/hour/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
nanomole/hour/milliliter
  Baseline (N=4, 5, 4) | 924.0 (1431) | 1481 (1165) | 367.0 (179.0)
  Change at Week 26 (N=4, 4, 4) | -76.0 (393.9) | -228 (692.7) | 94.75 (103.6)

17. Other Pre Specified Outcome: Change From Baseline in Neurofilament Proteins (NFP), Glial Fibrillary Acidic Protein (GFAP) and Tauprotein in Cerebrospinal Fluid (CSF) at Week 26
Time Frame: Baseline, Week 26
Population: ITT. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
nanogram/milliliter
  NFP: Baseline (N=4, 5, 4) | 5436 (3698) | 7848 (4510) | 12558 (3529)
  NFP: Change at Week 26 (N=4, 4, 4) | 1134 (8098) | -3505 (2553) | -4020 (9061)
  GFAP: Baseline (N=4, 5, 4) | 1758 (397.4) | 1014 (524.3) | 1415 (625.7)
  GFAP: Change at Week 26 (N=4, 4, 4) | 330.0 (380.3) | 402.5 (460.5) | 502.5 (285.4)
  Tauprotein: Baseline (N=4, 5, 4) | 1148 (143.4) | 1014 (530.9) | 1610 (543.4)
  Tauprotein: Change at Week 26 (N=4, 4, 4) | -288 (692.3) | -273 (228.7) | -118 (907.6)

18. Other Pre Specified Outcome: Change From Baseline in Amplitude at Week 26
Description: Abbreviations: MN=Median Nerve; PN=Peroneal Nerve; SN=Sural Nerve; Dig.=Digit; APB=abductor pollicis brevis; EDB=extensor digitorum brevis.
Time Frame: Baseline, Week 26
Population: ITT. Here, "N" signifies the number of participants who were evaluable for the respective category.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
millivolts
  MN, Wrist-APB: Baseline (N=4,5,4) | 5.63 (1.73) | 7.88 (2.20) | 4.30 (1.05)
  MN, Wrist-APB: Change at Week 26 (N=4,4,4) | 0.00 (2.84) | 0.65 (0.74) | -0.35 (1.66)
  MN, Elbow-APB: Baseline (N=4,5,4) | 3.85 (1.23) | 6.34 (2.71) | 2.65 (0.60)
  MN, Elbow-APB: Change at Week 26 (N=4,4,4) | 0.15 (2.05) | 0.33 (0.57) | -0.55 (0.65)
  MN, Dig. II Wrist: Baseline (N=4,5,4) | 2.68 (1.30) | 11.64 (14.89) | 1.78 (0.83)
  MN, Dig. II Wrist: Change at Week 26 (N=4,4,4) | -0.32 (1.00) | 3.53 (6.60) | -0.93 (0.85)
  PN, Ankle EDB: Baseline (N=4,4,4) | 1.85 (0.91) | 5.40 (2.55) | 1.30 (0.68)
  PN, Ankle EDB: Change at Week 26 (N=4,3,4) | -0.72 (1.66) | -0.43 (1.56) | 0.08 (0.96)
  PN, FH EDB: Baseline (N=4,4,4) | 2.43 (1.80) | 4.98 (2.95) | 0.95 (0.74)
  PN, FH EDB: Change at Week 26 (N=4,3,4) | -1.68 (2.06) | -0.63 (1.46) | 0.16 (0.75)
  SN, Sensory L LM - MC: Baseline (N=4,4,4) | 5.25 (6.31) | 41.18 (51.50) | 1.65 (2.28)
  SN, Sensory L LM - MC: Change at Week 26 (N=4,3,4) | -2.45 (4.18) | 0.53 (21.75) | -0.78 (2.34)
  SN, Sensory R LM - MC: Baseline (N=4,4,4) | 5.35 (5.45) | 50.05 (56.13) | 1.73 (2.01)
  SN, Sensory R LM - MC: Change at Week 26 (N=0,0,0) | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported. | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported. | NA (NA) — Since there were no participants evaluable for SN, Sensory R LM - MC category at Week 26, data could not be reported.

19. Primary Outcome: Maximum Plasma Drug Concentration (Cmax) of Recombinant Human Arylsulphatase A (rhASA)
Time Frame: Pre-dose and post-dose at 20, 40, 90 minutes, 3, 6 and 8 hours on Day 0, 40 minutes post-dose at Week 4, Pre-dose and post-dose at 20, 40, 90 minutes, 3, 6 and 8 hours at Week 8
Population: Due to quick disappearance of rhASA from plasma, rhASA levels were not possible to report.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

20. Primary Outcome: Arylsulfatase A (ASA) Activity in Leukocytes
Time Frame: Pre-dose and post-dose at 24 hours on Day 0 and at Weeks 8 and 26
Population: Data were not available to report as ASA activity in leukocytes was presented graphically, as per planned analysis.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

21. Other Pre Specified Outcome: Physical Examination Results
Description: Physical examination included general appearance, skin, head, ears, eyes, nose and throat, lymph nodes, heart, lungs, abdomen, extremities/joints, hip, neurological, mental status and, if appropriate, breasts, external genitalia, pelvic and rectal, and in addition weight, height and head circumference were recorded.
Time Frame: Baseline up to Week 26
Population: Physical examination results were not summarized since data were collected in participant's listing only as planned.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: From study drug administration up to Week 28 until evaluation (when last cohort had 26-week evaluation and data management performed within 4 weeks)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=5) | Cohort 3 (N=4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=5) | Cohort 3 (N=4)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (6) | 2 (3)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Type III immune complex mediated reaction (Immune system disorders) | 2 (12) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Drug specific antibody present (Investigations) | 2 (2) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mutism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
ASA activity in leukocytes could not be included in basic results format as the results were presented graphically. Due to quick disappearance of rhASA from plasma, rhASA levels were not possible to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.